CLINICAL TRIAL: NCT04597164
Title: Double Plasma Molecular Adsorption System With Sequential Low-Dose Plasma Exchange in Patients With Hepatitis B Virus-Related Acute-on-Chronic Liver Failure: A Prospective Cohort Study
Brief Title: Combination of DPMAS and Low Volume PE for Patients With HBV Related ACLF
Status: Recruiting | Type: Observational
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Liang Peng, Professor, Third Affiliated Hospital, Sun Yat-Sen University
Other Study IDs: PL13
Record Dates: First submitted 2020-10-08; First posted 2020-10-22 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Hepatitis B, Chronic; Acute-On-Chronic Liver Failure
Keywords: hepatitis b virus; acute-on-chronic liver failure; double plasma molecular adsorption system; plasma exchange
MeSH Terms: conditions — Hepatitis B, Chronic; Acute-On-Chronic Liver Failure; Hepatitis B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Artificial liver support system group: 100 patients in this group will receive treatment of double plasma molecular adsorption system, low volume plasma exchange, and comprehensive internal medical treatment
  Interventions: Other: Artificial liver support system
- Comprehensive medical treatment group: 100 patients in this group will receive comprehensive internal medical treatment.

INTERVENTIONS:
Other: Artificial liver support system — Patients will receive treatment of double plasma molecular adsorption system (DPMAS) and low volume plasma exchange (PE) for three times, and comprehensive internal medical treatment. The volume of plasma adsorption in DPMAS is 5000~6000 millilitre. The volume of fresh frozen plasma used in PE is 1000 millilitre.
  Groups: Artificial liver support system group

SUMMARY:
This study is to investigate investigate the safety and efficacy of Double plasma molecular adsorption system with sequential low-dose plasma exchange in treating hepatitis B virus-related acute-on-chronic liver failure.

DETAILED DESCRIPTION:
Hepatitis b virus (HBV) related acute-on-chronic liver failure (ACLF) is a serious condition with high mortality rate in China. But there still lacks of effective therapies in treatment of HBV related ACLF, except liver transplantation. Non-bioartificial liver support system treatments may be effective due to previous clinical data. Plasma exchange (PE) and double plasma molecular adsorption system (DPMAS) are two common ways in clinical practice. This study is to investigate the clinical efficacy and safety of combination treatment of DPMAS and low volume PE in patients with HBV related ACLF. This study will be completed in 6 medical center. Two hundred patients with HBV related ACLF enrolled in this study are divided into trial group (DPMAS, low volume PE, and comprehensive internal medical treatment) and control group (comprehensive internal medical treatment). Symptoms, signs, laboratory tests results, adverse events, mortality rates are recorded from treatment baseline to 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of chronic hepatitis b virus infection (positive hepatitis b surface antigen or positive hepatitis b virus DNA > 0.5 year);
2. Age from 18 to 65 years old;
3. Clinical diagnosis of liver failure (serum total bilirubin level > 10 times upper limit of normal; prothrombin time activity < 40% and ≥20%, or prothrombin time international ratio ≤ 2.6 and > 1.5);
4. Platelets > 50*10 E9/L.

Exclusion Criteria:

1. Other active liver diseases;
2. Hepatocellular carcinoma or other malignancy;
3. Pregnancy or lactation;
4. Human immunodeficiency virus infection or congenital immune deficiency diseases;
5. Severe diabetes, autoimmune diseases; unstable infarction due to cardio-cerebrovascular events;
6. Other important organ dysfunctions or transplantation;
7. Severe complications including severe infection, gastrointestinal bleeding, hepatic encephalopathy, hepatorenal syndrome;
8. Patients can not follow-up;
9. Investigator considering inappropriate.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This prospective study included patients diagnosed with HBV-ACLF at the Department of Infectious Diseases, the Third Affiliated Hospital of Sun Yat-sen University (Guangdong Province, China).
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-12-22 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Mortality or liver transplantation rate | 12 weeks
  Mortality or liver transplantation rate at 12-week follow-up.

SECONDARY OUTCOMES:
Model for end-stage liver disease (MELD) score variation | 12 weeks
  Variation of MELD score at 12 weeks after treatment. MELD score = 9.57 × loge(creatinine mg/dl) + 3.78 × loge(TBIL mg/dl) + 11.20 × loge(PT-INR) + 6.43.

CONTACTS AND LOCATIONS:
Overall Officials: Liang Peng, Doctor, Principal Investigator — Third Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
The study protocol, results and conclusions of this clinical trial will be published at academic conferences or in journals.
Supporting Information: Study Protocol, CSR
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Proposals should be directed to pliang@mail.sysu.edu.cn. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Derived] Xu W, Zhu S, Yang L, Li Z, Wu L, Zhang Y, Chen J, Deng Z, Luo Q, Peng L. Safety and efficacy of double plasma molecular adsorption system with sequential low-volume plasma exchange in intermediate-stage hepatitis B virus-related acute-on-chronic liver failure. J Med Virol. 2023 Mar;95(3):e28650. doi: 10.1002/jmv.28650. PMID 36897008
- [Derived] Xu W, Li Y, Wang L, Gao H, Chen J, Yuan J, Ouyang Y, Gao Y, Li J, Li X, Peng L. Efficacy and safety of combination treatment of double plasma molecular adsorption system and low volume plasma exchange for patients with hepatitis B virus related acute-on-chronic liver failure: a multicentre randomised controlled clinical trial. BMJ Open. 2021 Dec 14;11(12):e047690. doi: 10.1136/bmjopen-2020-047690. PMID 34907041